CLINICAL TRIAL: NCT06321185
Title: The Effects of Subcostal Transversus Abdominis Plane Block and Port-site Infiltration on the Quality of Recovery of Patients Undergoing Laparoscopic Cholecystectomy
Brief Title: Laparoscopic Cholecystectomy and Quality of Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Muserref Beril Dincer, Medical Doctor, Anesthesiologist, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024/177
Record Dates: First submitted 2024-03-14; First posted 2024-03-20 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Laparoscopic Cholecystectomy

STUDY DESIGN:
Intervention Model Description: The patients will be allocated randomly into three groups. Two groups will receive subcostal TAP block or port site local anesthetic infiltration, and the third group will not receive any intervention.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The subcostal TAP block and port-site infiltration will be applied after the patient has general anesthesia, so the patient will not know the allocated group. The healthcare providers who work in the ward and are responsible for the analgesic treatments will be blinded to the patient's group. The outcomes assessor who will question the QoR-15 scale at the 24th hour will also be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Subcostal TAP block (Active Comparator): Subcostal TAP block will be applied bilaterally with 20 ml 0.25% bupivacaine for each side.
  Interventions: Procedure: Subcostal TAP block
- Port site local anesthetic infiltration (Active Comparator): A total solution of 20 ml 0.25% bupivacaine will be infiltrated into the port sites before port placements.
  Interventions: Other: Port site local anesthetic infiltration
- Standard multimodal IV analgesia (Other): There will not be an intervention or local anesthetic administration.
  Interventions: Other: No intervention or local anesthetic administration

INTERVENTIONS:
Procedure: Subcostal TAP block — Subcostal TAP block will be applied after intubation and before surgery. A local anesthetic solution of 20 ml 0.25% bupivacaine for each side will be injected bilaterally between the rectus abdominis and transversus abdominis muscles along the oblique subcostal line. A multimodal routine IV analgesic regimen will be administered intraoperatively (1 gr paracetamol, 8 mg lornoxicam and 1mg/kg tramadol).
  Patients will receive a standard postoperative multimodal analgesia protocol comprising paracetamol and lornoxicam at the ward. Pain severity will be assessed with a Numeric Rating Scale (NRS) rated between 0 and 10; a rescue analgesic IV 50 mg tramadol will be applied when it is four or higher.
  Arms: Subcostal TAP block
Other: Port site local anesthetic infiltration — After intubation and before port placements, a solution of 20 ml 0.25% bupivacaine will be infiltrated into the laparoscopic port sites. A multimodal routine IV analgesic regimen will be administered intraoperatively (1 gr paracetamol, 8 mg lornoxicam and 1mg/kg tramadol).
  Patients will receive a standard postoperative multimodal analgesia protocol comprising paracetamol and lornoxicam at the ward. Pain severity will be assessed with a Numeric Rating Scale (NRS) rated between 0 and 10; a rescue analgesic IV 50 mg tramadol will be applied when it is four or higher.
  Arms: Port site local anesthetic infiltration
Other: No intervention or local anesthetic administration — There will not be an intervention or local anesthetic administration. A multimodal routine IV analgesic regimen will be administered intraoperatively (1 gr paracetamol, 8 mg lornoxicam and 1mg/kg tramadol).
  Patients will receive a standard postoperative multimodal analgesia protocol comprising paracetamol and lornoxicam at the ward. Pain severity will be assessed with a Numeric Rating Scale (NRS) rated between 0 and 10; a rescue analgesic IV 50 mg tramadol will be applied when it is four or higher.
  Arms: Standard multimodal IV analgesia

SUMMARY:
This clinical trial aims to compare the Quality of Recovery-15 (QoR-15) scale scores in three groups of patients undergoing laparoscopic cholecystectomy. The first group will be applied subcostal transversus abdominis plane (subcostal TAP) block, the second group will receive local anesthetic infiltration into port sites, and the third group will receive only IV analgesics.

DETAILED DESCRIPTION:
There are current approaches that search patients' perspectives to assess postoperative outcomes. In this regard, patient-centered outcomes are evaluated in clinical trials. It is recommended that patient comfort be assessed for short-term recovery after surgery. The Quality of Recovery-15 (QoR-15) scale is a defined patient comfort endpoint. This scale is a 15-item questionnaire that evaluates postoperative recovery as a patient-centered outcome. Each item is rated between 1 and 10, and the total score changes between 0 and 150. Improved recovery is associated with higher scores.

The subcostal transversus abdominis plane ( Subcostal TAP) block is used for analgesia in abdominal surgeries, including laparoscopic cholecystectomy. Local anesthetics are injected between the rectus abdominis and transversus abdominis muscles along the oblique subcostal line. Local anesthetic infiltration into the laparoscopic port sites is also used for analgesia in laparoscopic cholecystectomy.

The primary outcome of this study is to evaluate the effects of subcostal TAP block and port-site infiltration on the quality of recovery of patients undergoing laparoscopic cholecystectomy. Secondary outcomes are to evaluate Numerical Rating Scale (NRS) scores at time intervals, postoperative rescue analgesic requirement, total consumption of postoperative opioid analgesics, and presence of nausea and vomiting, for the postoperative 24 hours.

This study will be conducted as a prospective randomized clinical trial. The patients scheduled for elective laparoscopic cholecystectomy will be screened for enrollment in the study. After assessment for eligibility, the patients will be randomly allocated into three groups.

For the first group, a subcostal TAP block will be applied after intubation and before surgery. A local anesthetic solution of 20 ml 0.25% bupivacaine for each side will be injected bilaterally between the rectus abdominis and transversus abdominis muscles along the oblique subcostal line. For the second group, after intubation and before port placements, a solution of 20 ml 0.25% bupivacaine will be infiltrated into the laparoscopic port sites. The third group will not have an intervention or local anesthetic administration, and a multimodal routine IV analgesic regimen will be administered intraoperatively (1 gr paracetamol, 8 mg lornoxicam and 1mg/kg tramadol). This IV analgesic regimen will be applied to all patients included in the study. The patients will not know to which group they are allocated. Standard anesthesia protocol will be applied to all patients.

At the ward, patients will receive a standard postoperative multimodal analgesia protocol comprising paracetamol and lornoxicam. At the Numerical Rating Scale (NRS), pain is rated on a scale from 0 (no pain) to 10 (worst pain) and will be assessed at time intervals both at rest and during movement for postoperative 24 hours. A rescue analgesic IV 50 mg tramadol will be applied if it is four or higher. The healthcare provider will be blinded to which group the patient is in. All NRS scores, the requirement for rescue analgesics and total consumption, and the presence of nausea and vomiting for the postoperative 24 hours will be recorded by blind outcome assessors.

The Quality of Recovery-15 (QoR-15) scale will be evaluated before the surgery in the waiting area and at the postoperative 24th hour in the ward. The outcome assessor questioning QoR-15 will be blinded to which group the patient is allocated to.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective laparoscopic cholecystectomy
* Patients aged 18 to 80
* American Society of Anesthesiology (ASA) physical status I-II
* Signed informed consent

Exclusion Criteria:

* Patient refusal and inability to provide informed consent
* Known allergy to local anesthetics
* Severe kidney or liver disease
* Altered level of consciousness
* Inability to communicate due to language barrier
* Diagnosis of mental or psychiatric disorder
* Presence of coagulation disorder
* Contraindications to regional anesthesia
* Contraindications to any drug applying in the study
* Presence of coagulation disorder
* Chronic opioid intake
* Body mass index (BMI) ≥ 40 kg/m2
* History of alcohol or drug abuse
* Changed surgical technique from laparoscopic to open.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2024-03-25 (Actual); Primary Completion 2025-04-10 (Actual); Study Completion 2025-04-10 (Actual)

PRIMARY OUTCOMES:
Quality of Recovery-15 (QoR-15) scale | 24 hours
  Quality of Recovery-15 scale is a 15-item questionnaire that evaluates postoperative recovery as a patient-centered outcome. Each item is rated between 0 and 10, and the total score changes between 0 and 150. Improved recovery is associated with higher scores. Postoperative score at the 24th hour will be assessed as the primary outcome.

SECONDARY OUTCOMES:
Postoperative rescue analgesic requirement | 24 hours
  IV 50 mg tramadol will be administered as a rescue analgesic when patients Numerical Rating Scale (NRS) score is 4 and higher.
Consumption of postoperative opioid analgesics | 24 hours
  IV 50 mg tramadol will be administered when patients Numerical Rating Scale (NRS) score is 4 and higher. Total given dose of tramadol will be questioned.
Numerical Rating Scale (NRS) scores | 24 hours
  On the Numerical Rating Scale, pain is rated on a scale from 0 (no pain) to 10 (worst pain) and will be assessed at time intervals both at rest and during movement. Higher scores are related to severe pain.
Postoperative nausea and vomiting | 24 hours
  The presence of nausea and vomiting will be recorded postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Muserref B Dincer, Principal Investigator — Istanbul University Istanbul Medical Faculty
Locations (1):
- Istanbul University Istanbul Medical Faculty, Department of Anesthesiology and Reanimation, Istanbul, Fatih, Turkey (Türkiye)